CLINICAL TRIAL: NCT03971344
Title: Impact of Serious Pediatric Illness on Parent and Sibling Health
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Cigna Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: FP00024612
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Family Members of: Newborns Extremely Premature; Family Members of: New Pediatric Oncology Patients; Family Members of: Critical Congenital Heart Defect Patients; Family Members of: Children Severe Neurological Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Family members of newborns extremely premature: Parents and siblings (if any) of infants born at 30 weeks gestational age or less, or with a birthweight less than 1500 grams.
- Family members of new pediatric oncology patients: Parents and siblings (if any) of patients with new onset (not relapses) pediatric oncologic diagnoses including liquid, solid, and brain cancer.
- Family members of critical congenital heart defect patients: Parents and siblings (if any) of newborns with critical congenital heart defects who typically undergo surgery by 12 months of life.
- Family members of children with severe neurological impairment: Parents and siblings (if any) of patients with severe neurologic impairments, associated with substantial functional impairment, relentless progressive deterioration, or substantially shortened life-spans.

SUMMARY:
To estimate the impact of having a child with serious illness (SI) on the health and healthcare of other members of the child's family.

DETAILED DESCRIPTION:
Although standard pediatric practice, when caring for a child with serious illness, is to provide support to the child's parents and any siblings, little quantitative information exists regarding what could be considered the "collateral impact" on other family members of having a child with serious illness in the family. This study seeks to provide such information, using existing claims data from the health insurance company, Cigna, to identify children with serious illness and then examining the health and health care of their family members. The investigators hypothesize that, compared to control families without a sick child, parents and siblings of children with serious pediatric illness (SPI) will have more new mental and physical health diagnoses, more new prescriptions, increased levels of Emergency Department (ED) and acute care services, and reduced levels of use of recommended chronic disease management for pre-existing conditions and of preventative services.

ELIGIBILITY:
Inclusion Criteria:

* Cigna customers as follows:

  1. Neonatal Intensive Care Unit (NICU) cohort: infants born at 30 weeks gestational age or less, or with a birthweight less than 1500 grams.
  2. Critical Congenital Heart Disease (CCHD) cohort: Newborns with critical congenital heart defects who undergo surgery by 12 months of life.
  3. Oncology cohort: Patients with new onset (not relapses) pediatric oncologic diagnoses including liquid, solid, and brain cancer.
  4. Severe Neurological Impairment (NI) cohort: Patients with severe neurologic impairments, associated with substantial functional impairment, relentless progressive deterioration, or substantially shortened life-spans.
* For each index patient in a particular SPI cohort, Investigators randomly identified up to four children of the same ages as the index patient but who do not have the specific SPI. The matching by age was as follows: in months if < 3 years; and in years if age > or = 3 years. Cigna then identified all family members, using both definitions of "family members" described above.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: See Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 161000 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
New mental health diagnoses among parents | 3 years
  Outcome will be assessed based on diagnoses in de-identified claims data
New mental health diagnoses among siblings | 3 years
  Outcome will be assessed based on diagnoses in de-identified claims data
New physical health diagnoses among parents | 3 years
  Outcome will be assessed based on diagnoses in de-identified claims data
New physical health diagnoses among siblings | 3 years
  Outcome will be assessed based on diagnoses in de-identified claims data
New mental health prescriptions among parents | 3 years
  Outcome will be assessed based on prescription data in de-identified claims data
New mental health prescriptions among siblings | 3 years
  Outcome will be assessed based on prescription data in de-identified claims data
New physical health prescriptions among parents | 3 years
  Outcome will be assessed based on prescription data in de-identified claims data
New physical health prescriptions among siblings | 3 years
  Outcome will be assessed based on prescription data in de-identified claims data

SECONDARY OUTCOMES:
Emergency department usage among parents | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Emergency department usage among siblings | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Ambulatory care usage among parents | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Ambulatory care usage among siblings | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Hospitalizations among parents | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Hospitalizations among siblings | 3 years
  Outcome will be assessed based on encounter data in de-identified claims data
Adherence to chronic disease management standards among parents | 3 years
  Outcome will be assessed based on data in de-identified claims data
Receipt of well-child visit and childhood immunizations among siblings | 3 years
  Outcome will be assessed based on data in de-identified claims data

CONTACTS AND LOCATIONS:
Overall Officials: Chris Feudtner, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States